CLINICAL TRIAL: NCT06357000
Title: Association Between Time From PCI to Cancer Surgery and Cardiovascular and Oncologic Outcomes
Brief Title: Time From PCI to Cancer Surgery and Cardiovascular and Oncologic Outcomes
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: Time from PCI to surgery
Record Dates: First submitted 2024-04-03; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Cancer
Keywords: Time; Percutaneous coronary intervention; Cancer surgery
MeSH Terms: conditions — Coronary Artery Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time between the dates of PCI and cancer surgery <12 months: Time between the dates of PCI and cancer surgery <12 months
- time between the dates of PCI and cancer surgery ≥12 months: time between the dates of PCI and cancer surgery ≥12 months

SUMMARY:
To evaluate the association between time from PCI to cancer surgery and cardiovascular and oncologic outcomes in early-stage cancer patients, A retrospective, population-based cohort study was conducted using data from the Korean National Health Insurance Service (K-NHIS) database.

DETAILED DESCRIPTION:
Early-stage-cancer patients with a history of PCI who underwent cancer surgery (N = 3621) were included. The patients were divided into two groups based on the time between the dates of PCI and cancer surgery (<12 months and ≥12 months). Patients were stratified into early-surgery and late-surgery, defined as patients who underwent surgery ≥1 and <1 month after cancer diagnosis. Outcomes included bleeding, spontaneous myocardial infarction (MI), repeat revascularization, cancer recurrence, and death.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged ≥18 years who were diagnosed with cancer and underwent cancer surgery within 1 year following diagnosis.
* patients who underwent PCI (procedure code: M6551-M6572, O1640-O1649, OA640-OA649) prior to the cancer surgery

Exclusion Criteria:

* participants who received neoadjuvant or adjuvant treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early-stage cancer patients who underwent PCI before the cancer surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3621 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Occurence of Bleeding | up to 5 years
  Bleeding requiring transfusion was defined by the transfusion codes (X2021, X2022, X2031, X2032, X2091, X2092, X2111, X2112, X2131, X2132).

SECONDARY OUTCOMES:
Occurence of Spontaneous myocardial infarction | up to 5 years
  Spontaneous myocardial infarction (MI) was defined as hospitalization for MI (ICD-10 codes I21 and I22)
Occurence of Repeat revascularization | up to 5 years
  Repeat revascularization was defined as the presence of a procedure code after cancer surgery.
Occurence of Cancer recurrence | up to 5 years
  Cancer recurrence was defined as the presence of chemotherapy and/or radiation therapy that began more than 6 months after surgery completion.
Occurence of All cause death | up to 5 years
  Vital status was obtained from death certification collected by Statistics Korea at the Ministry of Strategy and Finance of South Korea.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi KH, Lee J, Lee J, Cho J, Kang D, Kim HK. Association Between Time From Percutaneous Coronary Intervention to Cancer Surgery and Cardiovascular and Oncological Outcomes. J Am Heart Assoc. 2025 May 6;14(9):e038569. doi: 10.1161/JAHA.124.038569. Epub 2025 Apr 16. PMID 40240888